CLINICAL TRIAL: NCT02765451
Title: Randomized Trial Evaluating Intervention of the Cancéropôle Nord-Ouest in the Development of Clinical Research in Non-Academic Health Institutions (ERNU)
Brief Title: Study Evaluating Intervention in the Development of Clinical Research in Non-Academic Health Institution (ERNU)
Acronym: ERNU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre de traitement des données du Cancéropôle Nord-Ouest, Centre F. BACLESSE, Caen, France (Unknown); Institut National de la Santé et de la Recherche Médical (INSERM) 1086 (Pr Guy LAUNOY) Centre F. BACLESSE, Caen, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RNI 2015-05-DR-BARBARE
Record Dates: First submitted 2016-04-27; First posted 2016-05-06 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Clinical Research; Cancer
Keywords: non-academic; health institution; development; clinical research; cancer; private hospital; public hospital; northwestern france; france; hospitals
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A : 1 year of intervention (Active Comparator): interventions of Cancéropôle Nord-Ouest during 1 year after an observational period of 2 years.
  Interventions: Behavioral: interventions of the Cancéropôle Nord-Ouest
- B : 2 years of intervention (Active Comparator): interventions of Cancéropôle Nord-Ouest during 2 years after an observational period of 1 year.
  Interventions: Behavioral: interventions of the Cancéropôle Nord-Ouest

INTERVENTIONS:
Behavioral: interventions of the Cancéropôle Nord-Ouest — During the time defined by the randomization, the Cancéropôle Nord-Ouest offers to help to develop a clinical research activities in the centers. The various aids are : Structuring clinical research at the local level, Support (strategy, logistics, technical, Data management, methodology), a portfolio of "straightforward" studies ( French National Cancer Institute, cooperative groups conducting cancer clinical research, New Project), Good Clinical Practice training, Clinical research technician, Others,.....

SUMMARY:
This study evaluates the interventions of the Cancéropôle Nord-Ouest in the development of clinical research in non-academic health institution. The randomization, in open label,determines the duration of the interventions. Half of participants will receive the interventions during 2 years, while the other half during 1 year.

DETAILED DESCRIPTION:
French National recommendations ask to increase the accessibility of patients to clinical trials. But this accessibility is far from the optimal care in non-university healthcare institutions (public and private hospital). These non-academic healthcare facilities support at national level about 60% of chemotherapy and 70% of radiotherapy, but only 17% of the inclusions in trials.

A dissociation exist between a care package guaranteed on quality criteria (criteria to obtain the capacity to treat the cancers in healthcare institution) distributed all over the country, and the research, mainly concentrated in few referral centers (University hospital and French Comprehensive Cancer Centers).

Clinical trials allow patients to have early access to new treatments, optimal and formalized information, and supported by physicians in connection with a strict protocol for patients included.

Several studies have shown the existence of geographical and socio-economic determinants for access to reference centers and for the duration of survival of cancer patients. In France, it was found that for patients with gastrointestinal cancer, the remoteness of the place of residence compared to the nearest referral center and a higher level of deprivation decreased the probability of being supported in a reference center.

The hypothesis of the ERNU study is that aid from the Cancéropole Nord-Ouest facilitates clinical research activity resulting in a significant development of inclusions in non-university centers of the french north-west inter-region with an influence on the social and geographical inequalities recruitment.

ELIGIBILITY:
Inclusion Criteria:

* French Health institutions of the Basse-Normandie, Haute-Normandie, Nord-Pas-de-Calais and Picardie.
* Health institutions non-academic public and private.
* Health institutions authorized to treat cancer.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2018-11-15 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Number of inclusions in clinical trials of patients | up to 2 years
  Measure the increase in inclusions in clinical trials of patients attending a Hospital or a private clinic "authorized to treat cancer" associated with a support provided by the Cancéropôle Nord-Ouest

SECONDARY OUTCOMES:
Reduction of social inequalities recruitment in clinical trials associated with the intervention of the Cancéropôle Nord-Ouest | up to 2 years
  assessment of the average of the reduction of social inequalities recruitment in clinical trial before and after the intervention of the Cancéropöle Nord-Ouest in each centers and in global. the social inequalities are calculated with the social and demographic tool developped by the french national institute of statistic and economic studies

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude BARBARE, MD, Study Director — Centre Hospitalier Universitaire Amiens Picardie
Locations (41):
- France (41):
  - Centre hospitalier d'Abbeville, Abbeville
  - Clinique de l'Europe, Amiens
  - Clinique Victor Pauchet, Amiens
  - Hopital Privé d'Arras, Arras
  - Centre hospitalier d'Arras, Arras
  - Centre de Radiothérapie de la Baie, Avranches
  - Centre Hospitalier de Bayeux, Bayeux
  - Clinique du Parc Saint Lazare, Beauvais
  - Centre hospitalier de Beauvais, Beauvais
  - Centre de Radiothérapie Pierre Curie, Beuvry
  - Centre Hospitalier de Béthune, Béthune
  - Centre Hospitalier de Boulogne sur Mer, Boulogne-sur-Mer
  - Centre de Radiothérapie Maurice TUBIANA, Caen
  - Polyclinique du Parc, Caen
  - Centre hospitalier de Calais, Calais
  - Centre Hospitalier de Cherbourg, Cherbourg
  - Centre hospitalier Compiègne-Noyon, Compiègne
  - Clinique Saint Côme, Compiègne
  - Clinique de Flandre, Coudekerque-Branche
  - Centre hospitalier Creil-Senlis, Creil
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Centre Hospitalier intercommunal Eure-Seine, Évreux
  - Centre hospitalier de Flers, Flers
  - Centre Hospitalier de Granville, Granville
  - Centre Hospitalier d'Hazebrouck, Hazebrouck
  - Centre hospitalier de Saint Omer, Helfaut
  - Centre hospitalier de Laon, Laon
  - Centre Hospitalier du Havre, Le Havre
  - Centre Hospitalier de Lens, Lens
  - Centre de radiuothérapie Bourgogne, Lille
  - Centre Hospitalier d'arrondissement de Montreuil sur mer, Rang-du-Fliers
  - Clinique Mathilde, Rouen
  - Centre Hospitalier intercommunal d'Elbeuf-Louvier, Saint-Aubin-lès-Elbeuf
  - Clinique les Aubépines, Saint-Aubin-sur-Scie
  - Clinique de la Baie, Saint-Martin-des-Champs
  - Clinique de Saint-Omer, Saint-Omer
  - Clinique Saint Claude, Saint-Quentin
  - Centre hospitalier de Saint Quentin, Saint-Quentin
  - Centre hospitalier de Soissons, Soissons
  - Centre Hospitalier de Tourcoing, Tourcoing
  - Centre hospitalier de Valenciennes, Valenciennes